CLINICAL TRIAL: NCT05076487
Title: Effects of Episodic Food Insecurity on Psychological and Physiological Responses in African American Women With Obesity
Brief Title: Effects of Episodic Food Insecurity in African American Women With Obesity
Acronym: RESPONSES
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Candice A. Myers, Ph.D., Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2021-022
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Obesity; Food Insecurity
Keywords: Food Insecurity; Stress; Body Weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African American Women with Food Security: 30 African American women with obesity who are food secure
- African American Women with Food Insecurity: 30 African American women with obesity who are food insecure

SUMMARY:
The objective of this exploratory/developmental study is to investigate the episodic nature of food insecurity as a stressor via responses in body weight and psychological and physiological parameters longitudinally. Sixty African American women with obesity will be enrolled. Pennington Biomedical Research Center will coordinate this longitudinal study and measure 1) daily body weight remotely over 22 weeks and 2) psychological and physiological parameters via clinic assessments at the beginning and end of 22 weeks as well as assess episodes of food insecurity and stress on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* willing to provide written informed consent
* female
* self-reported race of African American or more than one race in which African American is identified
* 18 to 65 years of age
* BMI 30 to 50 kg/m2
* reported income ≤ 250% of the federal poverty level
* ability to complete questionnaires in English
* willing to archive blood and urine samples
* willing to fast for a minimum of 8-10 hours prior to clinic visits

Exclusion Criteria:

* male
* self-reported race other than African American or more than one race in which African America is not identified
* reported income > 250% of the federal poverty level
* given birth within the past 6 months, currently pregnant, or plans to become pregnant within 6 months
* currently breastfeeding
* currently participating in a weight loss program
* current use of prescription or OTC medication specifically for weight loss
* recent weight loss (+/-5% weight change in last 6 months by self-report). If ppt is on a prescription medication that impacts weight but meets weight stability criteria (+/-5% weight change in last 6 months by self-report), ppt will be deemed eligible
* past bariatric surgery within the past 5 years or plans for bariatric surgery within 3 months
* active cancer or cancer treatment
* serious digestive disorders that significantly alter metabolism and weight (like uncontrolled inflammatory bowel disease)
* other conditions that affect metabolism or body weight
* current diagnosis and active treatment for alcoholism or other illicit drugs of abuse
* uncontrolled significant thyroid disorder (controlled = 6 months of medication)
* uncontrolled significant diabetes (FBS >250) or hypertension (BP >180/100)
* current diagnosis or treatment for heart failure
* serious psychiatric illness, including bipolar disorder and schizophrenia
* current or recent diagnosis (within last 5 years) of an eating disorder
* persons who weigh more than 380 pounds (due to scale)
* not willing to be able to re-contacted
* are unable to utilize devices and/or applications as required for study participation
* have another member of the household (same address) that is a participant in RESPONSES
* other conditions that affect metabolism or body weight as determined by the PIs and MI
* presence of any cognitive, psychiatric, behavioral, or medical disorder that, in the opinion of the PIs or MI may interfere with study participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African American women aged 18-65 with obesity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Body weight | 22 weeks
  Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Candice A Myers, PhD, Principal Investigator — Pennington Biomedical Research; John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research
Locations (1):
- Pennington Biomedical Research, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Myers CA, Beyl RA, Hsia DS, Harris MN, Reed IJ, Eliser DD, Bagneris L, Apolzan JW. Effects of Episodic Food Insecurity on Psychological and Physiological Responses in African American Women With Obesity (RESPONSES): Protocol for a Longitudinal Observational Cohort Study. JMIR Res Protoc. 2023 Dec 20;12:e52193. doi: 10.2196/52193. PMID 38117554